CLINICAL TRIAL: NCT04962659
Title: Telehealth Mindfulness-Based Music and Songwriting for Parents of Children With Intellectual/Developmental Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Endowment for the Arts, United States (U.S. Federal Agency)
Responsible Party: Principal Investigator, Miriam Lense, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18632783820
Record Dates: First submitted 2021-06-25; First posted 2021-07-15 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Parents; Stress; Developmental Disability; Intellectual Disability; Autism Spectrum Disorder
MeSH Terms: conditions — Developmental Disabilities; Intellectual Disability; Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Music and Songwriting (Experimental): The Mindfulness-Based Music and Songwriting (MBMS) program involves up to 8 weekly sessions (~1 hour) delivered via telehealth.
  Interventions: Behavioral: Mindfulness-Based Music and Songwriting
- Business as Usual Control (No Intervention): No treatment control.

INTERVENTIONS:
Behavioral: Mindfulness-Based Music and Songwriting — The Mindfulness-Based Music and Songwriting (MBMS) program involves up to 8 weekly sessions (~1 hour each) delivered via telehealth. During sessions, the participant works with a therapist (e.g., board-certified music therapist) to learn and apply mindfulness practices via music-based meditations and mindful songwriting. Supported by the therapist, participants write two songs during the program.
  Arms: Mindfulness-Based Music and Songwriting

SUMMARY:
This is a pilot study of the feasibility and potential impact of a Mindfulness-Based Music and Songwriting program (delivered via telehealth) on stress and well-being in parents/caregivers of children with intellectual or developmental disabilities. Participants are randomized to participate in the mindfulness program or a business-as-usual control group.

DETAILED DESCRIPTION:
This is a pilot study of the feasibility and potential impact of a Mindfulness-Based Music and Songwriting program (delivered via telehealth) on stress and well-being in parents/caregivers of children with intellectual or developmental disabilities. Participants are randomized to participate in the mindfulness program or a business-as-usual control group.

During mindfulness sessions, parents/caregivers are supported by a therapist to learn and apply mindfulness practices through music-based meditations and songwriting. Participants write two songs during the program. Parents complete surveys throughout the program.

ELIGIBILITY:
Inclusion Criteria:

* Parent/caregiver of a child with an intellectual or developmental disability
* Parent speaks and reads fluent English
* Able to attend weekly telehealth/virtual sessions

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2022-08-16 (Actual)

PRIMARY OUTCOMES:
Perceived stress | Baseline to end of study (baseline, within 1-week post-intervention, 4-week follow-up)
  Changes in perceived stress (self report: Perceived Stress Scale; higher score is higher stress)
Parent depression | Baseline to end of study (baseline, within 1-week post-intervention, 4-week follow-up)
  Changes in parent depression (self report rating scale: Beck Depression Inventory-II; higher score is higher depressive symptoms)
Parent well-being | Baseline to end of study (baseline, within 1-week post-intervention, 4-week follow-up)
  Changes in parent well-being (self-report rating scale: Ryff's Well-Being Scale; higher score is higher well-being)
Parent mindfulness | Baseline to end of study (baseline, within 1-week post-intervention, 4-week follow-up)
  Changes in parent mindfulness (self-report: Freiburg Mindfulness Inventory; higher score is higher mindfulness)
Parent positive reappraisal | Baseline to end of study (baseline, within 1-week post-intervention, 4-week follow-up)
  Changes in parent positive reappraisal (self-report scale; higher score is higher use of reappraisal)
Parent anxiety | Baseline to end of study (baseline, within 1-week post-intervention, 4-week follow-up)
  Changes in parent anxiety (self report rating scale: Beck Anxiety Inventory; higher score is higher anxiety symptoms)

SECONDARY OUTCOMES:
Parent affect regulation to MBMS sessions | Immediately pre and immediately post intervention sessions
  Changes in parent momentary affect (positive and negative affect subscales from Positive and Negative Affect Schedule (PANAS)) collected around mindfulness sessions (MBMS group only) (higher scores reflect higher positive affect and higher negative affect on respective subscales)
Parent social connection to therapist at MBMS sessions | Immediately pre and immediately post intervention sessions
  Changes in parent social connection (Inclusion of Other in the Self (IoS) scale) to therapist collected around mindfulness sessions (MBMS group only) (higher scores reflect higher social connection)
Parent daily momentary affect | 8-weeks (baseline, mid-intervention, post-intervention)
  Changes in parent daily momentary affect (collected via ecological momentary assessment with the Positive and Negative Affect Schedule (PANAS)) (higher scores reflect higher positive affect and higher negative affect on respective subscales)

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No